CLINICAL TRIAL: NCT04680065
Title: Randomized, Double-Blind, Placebo-controlled Safety Study of Glial Cell Line-Derived Neurotrophic Factor Gene Transfer (AAV2-GDNF) in Multiple System Atrophy
Brief Title: GDNF Gene Therapy for Multiple System Atrophy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brain Neurotherapy Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSA-101
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Multiple System Atrophy
Keywords: MSA; Multiple System Atrophy; Neurotrophic factor; Growth factor; Glial cell line-derived neurotrophic factor; GDNF; AAV; Gene therapy
MeSH Terms: conditions — Multiple System Atrophy | interventions — salicylhydroxamic acid; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Up to 9 study participants meeting eligibility criteria will be randomized in a 2:1 fashion to receive either the investigational medicinal product or sham surgery in this Phase 1 trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental)
  Interventions: Biological: AAV2-GDNF gene therapy
- Placebo Surgery (Sham Comparator)
  Interventions: Procedure: Sham (Placebo) Surgery

INTERVENTIONS:
Biological: AAV2-GDNF gene therapy — Bilateral image-guided infusion of AAV2-GDNF into putamen, single dose
  Arms: Active Treatment
Procedure: Sham (Placebo) Surgery — Bilateral partial burr/twist holes without dural penetration
  Arms: Placebo Surgery

SUMMARY:
The objective of this randomized, double-blinded, placebo-controlled Phase 1 investigation is to evaluate the safety and potential clinical effect of AAV2-GDNF delivered to the putamen in subjects with either a possible or probable diagnosis of Multiple System Atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 35-75 years of age (inclusive)
* Clinical diagnosis of MSA, parkinsonian type with symptoms onset sporadic, progressive and > 30 years of age
* Less than 5 years from MSA parkinsonian diagnosis with expected survival more than 3 years
* Stable anti-parkinsonian medication regimen
* Ability to walk a distance of 25 feet with or without an assistive device

Exclusion Criteria:

* Presence of idiopathic Parkinson's disease (PD) or any PD-related mutation or other neurological diseases
* Presence of dementia, psychosis, substance abuse or poorly controlled depression
* Prior brain surgery (i.e., deep brain stimulator implantation) or other brain imaging abnormalities
* History of cancer or poorly controlled medical conditions that would increase surgical risk
* Received investigational agent within 12 weeks
* Inability to tolerate laying flat in an MRI and/or allergy to gadolinium

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of Treatment-Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE) assessed clinically by physical and neurological examinations | 3 years
  Number of TEAE and SAE's reported post-treatment.

SECONDARY OUTCOMES:
MSA symptoms/signs as assessed by the Unified Multiple System Atrophy Rating Scale (UMSARS) | 12 months
  Change from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) and compared to placebo. UMSARS total scores range from 0-104 points with higher scores indicating greater severity of impairment.
Change in striatal dopamine transporter binding as measured by [123-I] Ioflupane | 12 months
  Percent and absolute change in ratio of specific to non-specific binding of 123I FP-CIT to DaT from baseline and compared to placebo by Single Photon Emission Computed Tomography (SPECT) dopamine transporter (DaT) imaging
Change in the quality of life as measured by Multiple System Atrophy Quality of Life (MSA-QoL) | 12 months
  Change from baseline and compared to placebo in the Multiple System Atrophy Quality of Life (MSA-QoL) scale. MSA-QoL is a self-reported questionnaire that measures MSA impact in day to day activities. Scale consists of 40 items with a five response option format (0 - no problem to 4 extreme problem) and a "not applicable" response option.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California Irvine, Irvine, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - NYU Langone Health, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nurse Navigator Service for Potential Participants — https://mytomorro.ws/msa-101-gov